CLINICAL TRIAL: NCT03774446
Title: A Phase 2 Multicenter Study of Seliciclib (R-roscovitine) for Cushing Disease
Brief Title: Multicenter Study of Seliciclib (R-roscovitine) for Cushing Disease
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Shlomo Melmed, MD, Sr. Vice President of Academic Affairs, Cedars-Sinai Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro52406; FD-R-6106 (Other Grant/Funding Number: Food & Drug Administration)
Record Dates: First submitted 2018-11-06; First posted 2018-12-13 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Cushing Disease
Keywords: Cushing disease; R-roscovitine; Seliciclib
MeSH Terms: conditions — Pituitary ACTH Hypersecretion | interventions — Roscovitine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Seliciclib (Experimental): 80 mg each day oral seliciclib for 4 weeks
  Interventions: Drug: Seliciclib

INTERVENTIONS:
Drug: Seliciclib — Drug: Seliciclib
  Other Names: R-roscotivine

SUMMARY:
This phase 2 multicenter, open-label clinical trial will evaluate safety and efficacy of 4 weeks of oral seliciclib in patients with newly diagnosed, persistent, or recurrent Cushing disease.

Funding Source - FDA Office of Orphan Products Development (OOPD)

DETAILED DESCRIPTION:
This phase 2 multicenter, open-label clinical trial will evaluate safety and efficacy of oral seliciclib in patients with newly diagnosed, persistent, or recurrent Cushing disease. Up to 13 subjects will be treated with 80 mg each day for 4 weeks. The study will also evaluate effects of seliciclib on quality of life and clinical signs and symptoms of Cushing disease.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients at least 18 years old
* Patients with confirmed pituitary origin of excess adrenocorticotropic hormone (ACTH) production:

  * Persistent hypercortisolemia established by two consecutive 24-hour UFC assessment ≥1.5× the upper limit of normal
  * Normal or elevated ACTH levels
  * Pituitary adenoma (>1 cm) on MRI or inferior petrosal sinus sampling (IPSS) central to peripheral ACTH gradient >2 at baseline and >3 after CRH stimulation
  * Recurrent or persistent CD defined as pathologically confirmed resected pituitary ACTH-secreting tumor or IPSS central to peripheral ACTH gradient >2 at baseline and >3 after CRH stimulation, and 24h-UFC >ULN beyond post-surgical week 6
* Patients on medical treatment for Cushing disease. The following washout periods must be completed before screening assessments are performed:

  * Inhibitors of steroidogenesis: metyrapone, ketoconazole: 2 weeks; Levoketoconazole: 3 weeks; osilodrostat: 6 weeks
  * Somatostatin receptor ligand pasireotide: short-acting, 2 weeks; long-acting, 4 weeks
  * Progesterone receptor antagonist mifepristone: 2 weeks
  * Dopamine agonist cabergoline: 4 weeks
  * Patients treated with CYP3A or CYP2B6 strong inducers or inhibitors, including those listed below. Required washout time varies between drugs; minimum 5-6 times the half-life of the drug.

    * Strong CYP3A inducers: apalutamide, carbamazepine, enzalutamide, mitotane, phenytoin, rifampin, St. John's wort
    * Moderate CYP3A inducers: bosentan, efavirenz, etravirine, phenobarbital, primidone
    * Weak CYP3A inducers: armodafinil, modafinil, rufinamide
    * Strong CYP2B6 inducer: carbamazepine
    * Moderate CYP2B6 inducers: efavirenz, rifampin
    * Weak CYP2B6 inducers: nevirapine, ritonavir
    * Strong CYP3A inhibitors: boceprevir, cobicistat, danoprevir and ritonavir, elvitegravir and ritonavir, grapefruit juice, indinavir and ritonavir, itraconazole, ketoconazole, lopinavir and ritonavir, paritaprevir and ritonavir and (ombitasvir and/or dasabuvir), posaconazole, ritonavir, saquinavir and ritonavir, telaprevir, tipranavir and ritonavir, telithromycin, troleandomycin, voriconazole, clarithromycin, idelalisib, nefazodone, nelfinavir.
    * Moderate CYP3A inhibitors: aprepitant, ciprofloxacin, conivaptan, crizotinib, cyclosporine, diltiazem, dronedarone, erythromycin, fluconazole, fluvoxamine, imatinib, verapamil
    * Strong CYP2B6 inhibitor: ticlopidine

Exclusion criteria:

* Patients with compromised visual fields, and not stable for at least 6 months
* Patients with abutment or compression of the optic chiasm on MRI and normal visual fields
* Patients with Cushing's syndrome due to non-pituitary ACTH secretion
* Patients with hypercortisolism secondary to adrenal tumors or nodular (primary) bilateral adrenal hyperplasia
* Patients who have a known inherited syndrome as the cause for hormone over secretion (i.e., Carney Complex, McCune-Albright syndrome, Multiple endocrine neoplasia (MEN) 1
* Patients with a diagnosis of glucocorticoid-remedial aldosteronism (GRA)
* Patients with cyclic Cushing's syndrome defined by any measurement of UFC over the previous 1 months within normal range
* Patients with pseudo-Cushing's syndrome, i.e., non-autonomous hypercortisolism due to overactivation of the hypothalamic-pituitary-adrenal (HPA) axis in uncontrolled depression, anxiety, obsessive compulsive disorder, morbid obesity, alcoholism, and uncontrolled diabetes mellitus
* Patients who have undergone major surgery within 1 month prior to screening
* Patients with serum K+< 3.5 while on replacement treatment
* Diabetic patients whose blood glucose is poorly controlled as evidenced by HbA1C >8%
* Patients who have clinically significant impairment in cardiovascular function or are at risk thereof, as evidenced by congestive heart failure (NYHA Class III or IV), unstable angina, sustained ventricular tachycardia, clinically significant bradycardia, high grade atrioventricular (AV) block, history of acute MI less than one year prior to study entry
* Patients with liver disease or history of liver disease such as cirrhosis, chronic active hepatitis B and C, or chronic persistent hepatitis, or patients with abnormal alanine transferase (ALT) or aspartate aminotransferase (AST) at screening or patients with advanced liver fibrosis (≥10 kPa) on elastography at screening
* Patients with estimated glomerular filtration rate (eGFR) <45 mL/min/1.73 m2
* Patients not biochemically euthyroid
* Patients who have any current or prior medical condition that can interfere with the conduct of the study or the evaluation of its results, such as

  * History of immunocompromise, including a positive HIV test result (ELISA and Western blot). An HIV test will not be required, however, previous medical history will be reviewed
  * Presence of active or suspected acute or chronic uncontrolled infection
  * History of, or current alcohol misuse/abuse in the 12 month period prior to screening
* Female patients who are pregnant or lactating, or are of childbearing potential and not practicing a medically acceptable method of birth control. If a woman is participating in the trial then one form of contraception is sufficient (pill or diaphragm) and the partner should use a condom. If oral contraception is used in addition to condoms, the patient must have been practicing this method for at least two months prior to screening and must agree to continue the oral contraceptive throughout the course of the study and for 3 months after the study has ended. Male patients who are sexually active are required to use condoms during the study and for three months afterwards as a precautionary measure (available data do not suggest any increased reproductive risk with the study drugs)
* Patients who have participated in any clinical investigation with an investigational drug within 1 month prior to screening or patients who have previously been treated with seliciclib
* Patients with any ongoing or likely to require additional concomitant medical treatment to treat CD
* Patients who have received pituitary irradiation within the last 5 years prior to the baseline visit
* Patients who have been treated with radionuclide at any time prior to study entry
* Patients with known hypersensitivity to seliciclib
* Patients with a history of non-compliance to medical regimens or who are considered potentially unreliable or will be unable to complete the entire study
* Patients with hepatitis B surface antigen (HbsAg) positivity
* Patients with hepatitis C antibody (anti-HCV) positivity
* Patients with prolonged QTcF on screening electrocardiogram (QTcF >450 msec)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Estimated)
Dates: Start 2018-11-02 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Number of participants with a normalized 24-hour urinary free cortisol (UFC) at study completion | 4 weeks
Number of participants with UFC above the upper limit of normal (ULN) but reduced by ≥50% from baseline at study completion | 4 weeks

SECONDARY OUTCOMES:
Plasma adrenocorticotrophic hormone | Baseline and week 4
Salivary cortisol | Baseline and week 4
Serum cortisol | Baseline and week 4
Glycated hemoglobin (HbA1c) | Baseline and week 4
Fasting blood glucose | Baseline and week 4
Weight and height to report body mass index (BMI) in kg/m^2 | Baseline and week 4
Blood pressure | Baseline and week 4
Change on visual field exam | Baseline and week 4
Change in tumor size on pituitary MRI | Baseline and week 4
Change in quality of life measured using the CushingQOL questionnaire | Baseline and week 4
Number of treatment-emergent adverse events graded using the National Cancer Institute (NCI) Common Toxicity Criteria (CTC) version 4.0 | Baseline and week 4

CONTACTS AND LOCATIONS:
Overall Officials: Shlomo Melmed, MD, Principal Investigator — Cedars-Sinai Medical Center; Ning-Ai Liu, MD, PhD, Study Director — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

REFERENCES:
- [Background] Liu NA, Araki T, Cuevas-Ramos D, Hong J, Ben-Shlomo A, Tone Y, Tone M, Melmed S. Cyclin E-Mediated Human Proopiomelanocortin Regulation as a Therapeutic Target for Cushing Disease. J Clin Endocrinol Metab. 2015 Jul;100(7):2557-64. doi: 10.1210/jc.2015-1606. Epub 2015 May 5. PMID 25942479
- [Background] Liu NA, Jiang H, Ben-Shlomo A, Wawrowsky K, Fan XM, Lin S, Melmed S. Targeting zebrafish and murine pituitary corticotroph tumors with a cyclin-dependent kinase (CDK) inhibitor. Proc Natl Acad Sci U S A. 2011 May 17;108(20):8414-9. doi: 10.1073/pnas.1018091108. Epub 2011 May 2. PMID 21536883